CLINICAL TRIAL: NCT02672293
Title: Determining Oral Phosphate Tolerance Across the Spectrum of Glomerular Filtration Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Rachel Holden (Other)
Responsible Party: Sponsor-Investigator, Dr. Rachel Holden, Principal Investigator, Queen's University
Organization: Queen's University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Holden/White; Queen's University (Other: Queen's University)
Record Dates: First submitted 2013-01-16; First posted 2016-02-03 (Estimated); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — sodium phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phosphate (Experimental): 500 mg of oral phosphate is administered after an overnight fast.
  Interventions: Drug: Phoslax

INTERVENTIONS:
Drug: Phoslax — Oral sodium phosphate solution (monobasic sodium phosphate 2.4 g and dibasic sodium phosphate 0.9g / 5 mL).
  Other Names: Sodium Phosphate

SUMMARY:
Over 20 million people in North America (including 2 million Canadians) have chronic kidney disease. These individuals die from diseases of the heart and blood vessels more often than they need dialysis. This is due to hardening of the arteries caused by calcium deposits inside the blood vessel walls. These deposits damage the vessels, causing them to lose flexibility. This makes them unable to respond to the changing demands of the body, and eventually leads to blockages such as stroke and ultimately death.

High levels of phosphate in the blood have been consistently linked to the development of calcium deposits inside blood vessel walls. The kidney is the only organ in the body that can eliminate phosphate that is not required by the body. As kidney function becomes worse, body levels of phosphate increase. However, investigators do not know the time point in the course of kidney disease that problems begin in the way phosphate is eliminated into the urine by the kidneys. Investigators will test the response of the kidneys to a phosphate challenge taken by mouth in subjects who are having accurate measures of kidney function performed by a method called 'inulin clearance'.

The investigators believe that the results of this study will provide important information identifying when investigators should be concerned about body levels of phosphate increasing. This information may lead to changes in the way investigators treat patients by reducing the levels of phosphate in the diet at a much earlier time point then is presently recommended.

DETAILED DESCRIPTION:
Fractional excretion of phosphate will be measured pre- and 60 minutes and 120 minutes following an oral challenge of 500 mg of oral phosphate in a group of patients with gold standard measures of glomerular filtration rate.

ELIGIBILITY:
Inclusion Criteria:

* stable chronic kidney disease

Exclusion Criteria:

* unable/unwilling to give informed consent;
* pregnant or breast-feeding;
* known allergy to shellfish, iodine or inulin;
* have evidence of impaired bladder emptying defined as a post-void residual of greater than 20 ml.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-01; Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
Fractional excretion of phosphate | Change in fractional excretion of phosphate at 1 and 2 hours
  Fractional excretion of phosphate will be measured at baseline and at 1 and 2 hours following a standardized oral phosphate challenge

SECONDARY OUTCOMES:
Fibroblast growth factor-23 | Change in level of fibroblast growth factor 23 at 2 hours
  Biomarker of phosphate homeostasis
Vitamin D | Change in level of vitamin D and vitamin D metabolites at 2 hours
  Biomarker of phosphate homeostasis
klotho | Change in level of circulation kloth at 2 hours
  Biomarker of phosphate homeostasis

CONTACTS AND LOCATIONS:
Overall Officials: Rachel M Holden, MD, Study Chair — Queen's University
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No